CLINICAL TRIAL: NCT06270446
Title: Community Based Rehabilitation Model After Total Knee Replacement: A Pilot Study
Brief Title: Community Based Rehabilitation Model After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSRB 2019/01135
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Masking Description: Data analysis blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient (Other): Usual care, outpatient physiotherapy
  Interventions: Other: Outpatient physiotherapy
- CRC (Active Comparator): Community based physiotherapy
  Interventions: Other: Community based physiotherapy

INTERVENTIONS:
Other: Community based physiotherapy — Physiotherapy at community rehabilitation center
  Arms: CRC
Other: Outpatient physiotherapy — Physiotherapy at hospital
  Arms: Outpatient

SUMMARY:
To investigate the clinical efficacy of community-based early stage knee replacement rehabilitation program as compared with usual care in acute hospital outpatient clinic

DETAILED DESCRIPTION:
To investigate the clinical efficacy of community-based early stage knee replacement rehabilitation program as compared with usual care in acute hospital outpatient clinic

ELIGIBILITY:
Inclusion Criteria:

i) unilateral TKA; ii) age 55 years old and above; iii) able to engage in outpatient physiotherapy; iii) postoperative knee flexion ≥75° and knee extension ≤5°; iv) able to ambulate independently preoperatively.

Exclusion Criteria:

i) had revision TKA or fully constrained knee arthroplasty; ii) had knee replacement for indications other than osteoarthritis; iii) had post-operative complications during hospital stay; iv) were unable to participate due to cognitive impairment or language barriers; v) had acute spinal diseases or joint, muscle or systemic diseases affecting gait; iv) had comorbid health conditions that would prevent active participation (e.g. prior hemiplegic stroke, severe cardiorespiratory illnesses.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
TUG | 3 months
  TUG score
30 sec chair stand test | 3 months
  30 sec chair stand test score
Pain intensity | 3 months
  Pain intensity score

SECONDARY OUTCOMES:
Knee flexion and extension | 3 months
  Knee flexion and extension ROM
Passive range of motion | 3 months
  Passive range of motion ROM
Presence of lag | 3 months
  Presence of knee extensor lag

OTHER OUTCOMES:
OKS | 3 months
  Oxford knee score

CONTACTS AND LOCATIONS:
Overall Officials: Eng Chuan Neoh, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore